CLINICAL TRIAL: NCT04608110
Title: A Phase 1, Multi-center, Open-label, Uncontrolled, Dose-escalation Study to Evaluate the Pharmacokinetics of ASTX030 in Patients With Myelodysplastic Syndrome (MDS)
Brief Title: A Phase 1 Trial of ASTX030 in Patients With Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 418-102-00001
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacitidine + Cedazuridine (Experimental): Drug: Azacitidine
  Tablets or capsules for oral administration and powder for reconstitution to aqueous suspension for subcutaneous administration
  Drug: Cedazuridine
  Tablets for oral administration
  Interventions: Drug: ASTX030

INTERVENTIONS:
Drug: ASTX030 — In Cycle 1 (28 days per cycle), single dose oral azacitidine formulations will be administered on day -3, followed by subcutaneous (SC) azacitidine on day 1, oral azacitidine formulations and cedazuridine tablets on day 2-7; in Cycle 2 and onward, oral azacitidine formulations and cedazuridine tablets will be administered on day 1-7

SUMMARY:
The purpose of this study is to identify the doses of the oral azacitidine formulations and cedazuridine (CED) tablets which achieve a total AUC for AZA comparable to that for AZA injection at 75 mg/m2

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older
* Patients with a diagnosis of MDS (refractory anemia [RA], refractory anemia with ringed sideroblasts [RARS], refractory anemia with excess blasts [RAEB], refractory anemia with excess blasts in transformation [RAEB-T], or chronic myelomonocytic leukemia [CMML]) according to the French-American-British (FAB) classification Low-risk patients who fall under the risk category of low or intermediate-1 (Int-1) based on the International Prognostic Scoring System (IPSS) can be enrolled only if they are unlikely to respond to any other treatment or if they are currently being treated with azacytidine (AZA) injection
* Patients with an ECOG PS score of 0 or 1 or with an ECOG PS score of 2 due to primary disease-associated conditions
* Patients with adequate organ function as indicated below

  1. Hepatic function: All of the following criteria must be satisfied.

     * Total bilirubin ≤ 2.0 × upper limit of normal (ULN)
     * Aspartate aminotransferase (AST) ≤ 2.5 × ULN
     * Alanine aminotransferase (ALT) ≤ 2.5 × ULN
  2. Renal function: Either of the following criteria must be satisfied.

     * Serum creatinine ≤ 1.5 × ULN
     * Creatinine clearance or glomerular filtration rate ≥ 50 mL/min
  3. Respiratory function: percutaneous arterial oxygen saturation (SpO2) ≥ 90%
* Patients who are expected to survive for at least 3 months
* Patients who give written consent to participate in the trial using the informed consent form approved by the institutional review board

Exclusion Criteria:

* Patients who are unlikely to respond to AZA
* Patients who have received chemotherapy, hormone therapy, antibody therapy, radiotherapy, or other exploratory anti-cancer treatments for the primary disease within 3 weeks prior to the first administration of the investigational medicinal product (IMP)
* Patients who have used any other IMP or any privately imported medicine within 4 weeks prior to the first administration of IMP
* Patients with heart disease of Class 3 or 4 according to the New York Heart Association classification
* Patients with uncontrolled systemic disease or active infection
* Patients with uncontrolled gastric or duodenal ulcer
* Patients with prior or current interstitial lung disease
* Patients with a history of surgical gastrectomy
* Patients with life-threatening conditions/symptoms, multiple organ failure, or other factors (including laboratory abnormalities) that, in the opinion of the investigator, are likely to affect their safety or the absorption and metabolism of AZA and cedazuridine (CED), or influence the trial evaluation
* Patients with other malignancies (except appropriately treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma in situ; prostate or breast cancer stabilized by endocrine therapies; and malignancies that have not relapsed for at least 1 year since the last successful treatment)
* Patients who are positive for HIV antibody, HBV-DNA, or HCV antibody
* Patients with any ≥ Grade 2 AE (except alopecia) associated with prior treatment of the primary disease. However, the parameters defined in inclusion criterion above are excluded.
* Patients who have undergone a highly invasive and extensive surgical procedure within 4 weeks prior to the first administration of IMP
* Patients who previously underwent or plan on undergoing hematopoietic stem cell transplantation
* Patients with a history of hypersensitivity to the active ingredient or any excipient of IMP
* Patients who are, in the opinion of the investigator, at high risk for being unable to comply with the trial protocol because of mental disorders or other medical conditions (alcohol/substance abuse or addiction)
* Pregnant or nursing female patients, or female patients with a positive pregnancy test at screening. Nursing patients cannot participate in the trial even if they discontinue breastfeeding. Female patients must undergo a pregnancy test to confirm that they are not pregnant at screening. However, a pregnancy test is not necessary for female patients without childbearing potential (ie, patients with a history of bilateral oophorectomy or hysterectomy or who have been postmenopausal for at least 12 months except for cases where menopause could be due to the effect of antineoplastic treatment).
* Sexually active males (except those with a history of bilateral orchiectomy) or females of childbearing potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 3 months (males) and 6 months (females) after the last dose of IMP. If birth control is employed, 2 of the following precautions must be used: vasectomy, tubal ligation, intrauterine device, oral contraceptive, and condom (all methods approved or certified in Japan)
* Patients who, in the opinion of the investigator, are otherwise ineligible to participate in the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
• AUC ratio of AZA after administration of oral azacitidine formultions in combination with CED tablets compared with subcutaneous (SC) administration of AZA injection | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (10):
- Japan (10):
  - Nippon Medical School Hospital, Bunkyō City
  - Fukushima Medical University Hospital, Fukushima
  - Saitama Medical University Hospital, Iruma
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Osaka City General Hospital, Osaka
  - Kindai University Hospital, Sakai
  - NTT Medical Center Tokyo, Shinagawa-Ku
  - Tokyo Medical University Hospital, Shinjuku-Ku
  - Yamagata University Hospital, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.